CLINICAL TRIAL: NCT01622881
Title: Analgesic Efficacy of Nefopam in Patients Undergoing Kidney Transplantation : Randomized Controlled Study
Brief Title: Analgesic Efficacy of Nefopam in Patients Undergoing Kidney Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, So Yeon Kim, Clinical assistant professor, Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2012-0173
Record Dates: First submitted 2012-06-13; First posted 2012-06-19 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Saline Solution; Nefopam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nefopam (Active Comparator)
  Interventions: Drug: Nefopam
- Control (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Normal saline — Normal saline 200mL : the infusion of 4mL/hr for post-operative 48 hours
  Arms: Control
Drug: Nefopam — Nefopam 160mg (16 mL) mixed to normal saline 184 mL : the infusion of 4mL/hr for post-operative 48 hours
  Arms: Nefopam

SUMMARY:
The investigators examined the efficacy of nefopam in patients undergoing kidney transplantation.

DETAILED DESCRIPTION:
Drug combination are frequently used to relieve postoperative pain. Nefopam can inhibit serotonin, dopamine, and norepinephrine reuptake through central mechanisms. Several studies have demonstrated analgesic efficacy of nefopam in the postoperative period. The purpose of this study is to ascertain the analgesic effect and tolerance of intravenous nefopam in combination with fentanyl based patient-controlled analgesia after kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* elective living donor kidney transplantation

Exclusion Criteria:

* pre-operative tachycardia (> 100bpm)
* liver dysfunction
* severe cardiac disease
* body mass index ≥ 30 kg/m2
* drug allergy

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Fentanyl consumption by patient-controlled analgesia | 48 hours
Numerical rating score of pain | 48 hours

SECONDARY OUTCOMES:
The number of patients who had side effects (e.g. nausea, vomiting, dizziness, headache, confusion, tachycardia) | 48 hours
Early postoperative graft function | until discharge
  serum creatinine, estimated glomerular filtration rate, delayed graft function defined as the need for dialysis within 1 week after surgery, acute rejection episodes included both biopsy-proven and clinically suspected acute rejection

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea